CLINICAL TRIAL: NCT04493333
Title: Comparison of Vaginal Dehydroepiandrosterone (DHEA) to Control for Treatment of Vaginal Symptoms in Postmenopausal Breast Cancer Survivors on Aromatase Inhibitors: A Phase II Randomized Trial
Brief Title: Vaginal Dehydroepiandrosterone (DHEA) in Postmenopausal Breast Cancer Survivors on Aromatase Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment/enrollment
Sponsor: University of Arkansas (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 239531
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Vaginal Atrophy; Postmenopausal Symptoms; Breast Cancer Female; Long-term Survivors
Keywords: Postmenopausal; Breast Cancer Survivor; Vaginal
MeSH Terms: interventions — Dehydroepiandrosterone; Replens

STUDY DESIGN:
Intervention Model Description: Subjects are randomly assigned to the Intrarosa® or Replens™ arm by a 1:1 ratio. Subjects randomized to the Intrarosa® arm will use 6.5 mg daily for 12 weeks (±1 week). Subjects randomized to the Replens™ arm will use a vaginal applicator two times per week for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: The cytologist's reading specimens will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaginal DHEA (Experimental): Vaginal insert with 6.5 mg vaginal DHEA self-administered once daily at bedtime for 12 weeks
  Interventions: Drug: Vaginal Dehydroepiandrosterone
- Vaginal Polycarbophil Moisturizer (Active Comparator): Prefilled vaginal applicator with 2.5 g of polycarbophil vaginal moisturizing gel, self-administered two times per week at night for 12 weeks
  Interventions: Combination Product: Vaginal Polycarbophil Moisturizer

INTERVENTIONS:
Drug: Vaginal Dehydroepiandrosterone — This is a vaginally administered suppository steroid indicated for the treatment of moderate to severe dyspareunia, a frequent symptom of vulvovaginal atrophy due to menopause or genitourinary syndrome of menopause.
  Other Names: Intrarosa®; Vaginal DHEA; Prasterone
  Arms: Vaginal DHEA
Combination Product: Vaginal Polycarbophil Moisturizer — This is an FDA cleared, over-the-counter personal lubricant for vaginal application, intended to moisturize and lubricate, to enhance the ease and comfort of intimate sexual activity and supplement the body's natural lubrication. It is non-sterile, water-based, non-irritating, non-greasy, non-staining vaginal gel delivered as a long-lasting moisturizer for vaginal dryness.
  Other Names: Replens™
  Arms: Vaginal Polycarbophil Moisturizer

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of Intrarosa®, also known as Dehydroepiandrosterone (DHEA), and prasterone. By doing this study, the investigators hope to learn if Intrarosa® can improve vaginal discomfort. Participants will be assigned to one of two groups. One group will use Intrarosa® once a day. The other group will use Replens™ two times a week.

DETAILED DESCRIPTION:
This will be a two-armed, randomized Phase II trial. All study subjects will be asked to fill out a simple 5-question sexual functioning survey. If any concern about sexual functioning is noted, the subject will also be asked to fill out a more extensive Sexual functioning tool, to help determine which domain of sexual functioning is the most bothersome.

Subjects who complete the initial screening will be randomly assigned to the Intrarosa® or Replens™ arm by a 1:1 ratio. Subjects randomized to the Intrarosa® arm will use 6.5 mg daily for 12 weeks (±1 week). Subjects randomized to the Replens™ arm will use a vaginal applicator two times per week for 12 weeks.

At baseline and at 12 weeks, subjects will undergo a physical exam including clinical breast and gynecological exam. During gynecologic exams, the vaginal Potential of Hydrogen (pH) will be determined and a swab of vaginal epithelium sent for determination of the Vaginal Maturation Index (VMI) and Maturation Value (MV). These will be used as objective physiologic markers to determine the improvement in vaginal atrophy. The cytologist's reading specimens will be blinded.

Additionally, all study subjects will be asked to fill out questionnaires at baseline and again in 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients with a history of breast cancer who have completed primary treatment with curative intent, who have been on an aromatase inhibitors (AI) for at least 6 months
* Stage I-III, hormone receptor positive breast cancer regardless of human epidermal growth factor receptor 2 (HER2) status
* Postmenopause defined as 12 months of spontaneous amenorrhea, or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL (milli-international units per milliliter), or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy. FSH level will be documented on all subjects.
* Patients reporting any symptoms of vaginal dryness or dyspareunia as assessed by the Brief Sexual Symptom Checklist for Women (BSSC-W) or the Female Sexual Function Index (FSFI)
* No evidence of active malignant breast or gynecologic disease
* Absence of undiagnosed, persistent or recurring genital bleeding that has not been evaluated to determine the cause [6]
* No planned changes in AI during the study period
* Mammogram (if appropriate, as determined by the treating physician and will be documented) within 12 months of study entry
* Patients with documented normal Pap within 12 months of study entry

Exclusion Criteria:

* Use of any estrogen or progesterone depot-preparation drug or progestin implant in the last 6 months before study entry
* Use of any androgen or anabolic steroids in the last 6 months before study entry
* Use of any oral or transdermal hormonal products (estrogen, progestin, or DHEA) within the last 8 weeks prior to study entry; however, a subject can elect to wait for an 8-week washout period before study entry.
* Use of any vaginal or intrauterine hormonal products in the last 8 weeks; however, a subject can elect to wait for an 8-week washout before study entry.
* Use of any natural over the counter estrogenic products in the last 6 months; however, a subject can elect to wait for a 6-month washout before study entry.
* Concomitant vulvar and vaginal surgical or laser treatments
* Vaginal infection or confounding vulvar or active vaginal disease process
* Prior radiation to the pelvis or history of gynecologic cancer
* Inability to tolerate a vaginal/speculum exam
* Undiagnosed, persistent or recurring genital bleeding or other indication of active pelvic disease process that has not been evaluated [6]
* Clinically significant uncontrolled depression or severe psychiatric symptoms
* If subject has an established routine of inert vaginal lubricant use for routine or occasional relief of vulvar or vaginal symptoms prior to the study period, it may be continued during the study period along with the study drug.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Richard-Davis, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be identified in the UAMS CI and UAMS Women's Health clinics and from the CARTI Cancer Center, during routine clinic appointments by the provider or research staff. Potential research subjects may also contact the UAMS Cancer Institute's Clinical Trials Office regarding participation based on the information found within the IRB-approved DHEA flyer that is to be distributed amongst UAMS and the CARTI medical clinics.
Pre-assignment Details: Females of childbearing age and potential must have negative pregnancy test at screening. Any consented individuals who do not indicate sexual complaints on Question 1 of the BSSC-W at baseline will be considered a screen fail and will not complete the FSFI or continue in the study.
Groups:
- Intrarosa & Standard of Care Aromatase Inhibitor: Subjects randomized to the Intrarosa® arm will use 6.5 mg daily for 12 weeks (±1 week).
- Replens & Standard of Care Aromatase Inhibitor: Subjects randomized to the Replens™ arm will use a vaginal applicator two times per week for 12 weeks (±1 week).
Period: Overall Study
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Started | 5 | 3
Completed | 2 | 0
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Ineligible | 0 | 1
Not completed — Noncompliance | 2 | 1

BASELINE CHARACTERISTICS:
Population: Postmenopausal females between 18 and 70 with a history of breast cancer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (3.96) | 54.00 (15.39) | 56.38 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 8
Vaginal Maturation Index (VMI) [Mean (Standard Deviation); unit: Units on a scale] — VMI is a clinical measure of vaginal estrogenization, indicator of the degree of vaginal atrophy which is the end result of treatment with aromatase inhibitors that leads to vaginal dryness and dyspareunia. VMI is the proportional relationship of parabasal (P) cells to intermediate (I) and superficial (S) cells in the vaginal epithelium. VMI = 1.0 x %S + 0.5 x %I + 0.0 x %P cells, which is VMI=%S + (0.5 x %I) when simplified, potential range of 0-100. A VMI of 65-100 suggests a normal premenopausal environment, 50-64 indicates a moderate estrogenic effect, and <50 indicates atrophy.
  Units on a scale | 50.83 (16.65) | 36.67 (23.23) | 43.75 (19.67)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Vaginal Maturation Index (VMI) Response From Baseline to Week 12
Description: The change in the subject's calculated VMI from baseline to the end of treatment at 12 weeks (±1 week). VMI = 1.0 x %S + 0.5 x %I + 0.0 x %P cells, which is the same as VMI = %S + (0.5 x %I) when simplified. It has a potential range of 0-100. A VMI of 65-100 suggests a normal premenopausal environment, 50-64 indicates a moderate estrogenic effect, and < 50 indicates atrophy.
Time Frame: Baseline and 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 had VMI measured at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | -7.5 (24.75) |

2. Secondary Outcome: Difference in Vaginal pH From Baseline to Week 12
Description: Vaginal pH was used as an objective physiologic marker to determine the improvement in vaginal atrophy. pH is a measure of acidity and alkalinity and can range from 0 to 14, with 7 being neutral. Lower pH scores are acidic and higher pH scores are basic or alkaline. A normal healthy vaginal pH is 4.5. As the vaginal epithelium becomes thinner and more atrophic, the mucosa has less glycogen content and less lactobacilli to convert the glycogen into lactic acid, which results in an increase in the vaginal pH.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 had vaginal pH measured at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | -1.00 (2.83) |

3. Secondary Outcome: Difference in Dyspareunia Scores on the Brief Sexual Symptom Checklist for Women (BSSC-W) From Baseline to Week 12
Description: The Dyspareunia Score on the BSSC-W asks if there is a problem with pain during sex. A difference score of 0 indicated no change in whether it was a problem. The min and max are both 0 which makes the range also 0. Only 2 participants had week 12 scores. These scores were both 1. (So the min and max were 1 with the range being 0.) Of the baseline scores, these 2 participants both had scores of 1 again. (So the min and max for these 2 participants were both 1 with a range of 0.) If we include these 2 participants with the other 6 who have baseline dyspareunia scores on the BSSC-W, then 7 participants has a score of 1 and 1 participant had a score of 0. This would make the min, max, and range 0, 1, and 1 respectively. As for which value represents a better or worse outcome, 1 indicates presence of dyspareunia while 0 indicates absence of dyspareunia, so 1 is a worse outcome than 0. Subscales are not combined here to produce a total score.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 took the BSSC-W at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | 0.00 (0.00) |

4. Secondary Outcome: Difference in Vaginal Dryness Scores on the Brief Sexual Symptom Checklist for Women (BSSC-W) From Baseline to Week 12
Description: The min and the max are both 0 which make the range also 0. These were obtained from subtracting each participant's score at baseline from their score at week 12. Only 2 participants had week 12 scores. These scores were both 1. Of the baseline scores, these 2 participants both had scores of 1 again. If 2 participants with the other 6 have baseline dyspareunia scores on the BSSC-W, then 7 participants have a score of 1 and 1 participant had a score of 0. This would make the min, max, and range 0, 1, and 1 respectively. As for which value represents a better or worse outcome, 1 indicates presence of vaginal dryness (problem with decreased vaginal lubrication) while 0 indicates absence of vaginal dryness (or an absence of this problem of decreased vaginal lubrication), so 1 is a worse outcome than 0. Subscales are not combined here to produce a total score.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 took the BSSC-W at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | 0.00 (0.00) |

5. Secondary Outcome: Difference in Dyspareunia Subscale Scores on the Female Sexual Dysfunction Index (FSFI) From Baseline to Week 12
Description: The Dyspareunia Subscale Score on the Female Sexual Dysfunction Index ranges from 0-5 with higher scores indicating better sexual function, so less dyspareunia.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 took the FSFI at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | 2.20 (3.11) |

6. Secondary Outcome: Difference in Vaginal Dryness Subscale Scores on the Female Sexual Dysfunction Index (FSFI) From Baseline to Week 12
Description: The Vaginal Dryness (or Lubrication) Subscale Score on the Female Sexual Dysfunction Index ranges from 0-5 with higher scores indicating better sexual function, so more lubrication.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 took the FSFI at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale | 1.80 (2.55) |

7. Secondary Outcome: Difference in Quality of Life on the Quality of Life - Cancer Survivor Version (QOL-CSV) From Baseline to Week 12
Description: The Quality of Life - Cancer Survivor Version ranges from 0-10 with higher scores indicating a higher quality of life. T here are only 2 difference scores for each of the 4 subscales. The min, max, and ranges of these Well-Being Subscales: Physical -1.00, -0.62, and 0.38. Psychological -0.72, 0.94, and 1.67. Social 0.75, 1.25, and 0.50. Spiritual -1.57, 3.29, and 4.86. For Psychological the min, max, and range are 2.61, 6.83, and 4.22. For Social the min, max, and range are 2.63, 7.38, and 4.75. For Spiritual the min, max, and range are 4.43, 8.43, and 4.00. A negative difference score indicates a worsening of quality of life while a positive score indicates that qualify of life got better. Subscales were not combined here to produce a total score. For the baseline and week 12 scores on the QOL-CSV, higher scores mean higher quality of life.
Time Frame: 12 weeks (±1 week)
Population: Out of 8 participants assigned to a treatment arm, only 2 took the QOL-CSV at both the baseline and 12-week visits.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
Number analyzed (Participants) | 2 | 0
Units on a scale
  QOL-CSV Physical Well-Being Subscale | -0.81 (0.27) |
  QOL-CSV Psychological Well-Being Subscale | 0.11 (1.18) |
  QOL-CSV Social Well-Being Subscale | 1.00 (0.35) |
  QOL-CSV Spiritual Well-Being Subscale | 0.86 (3.43) |

ADVERSE EVENTS:
Time Frame: 12 weeks (+/- 1 week)
Description: AEs are to be reported in a routine fashion at scheduled times during the trial. Certain AEs must be reported in an expedited fashion to allow for timely monitoring of subject safety and care.
Arm/Group | Intrarosa & Standard of Care Aromatase Inhibitor | Replens & Standard of Care Aromatase Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrarosa & Standard of Care Aromatase Inhibitor (N=5) | Replens & Standard of Care Aromatase Inhibitor (N=3)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Burning with vaginal Intrarosa application (General disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (3) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other, specify: Vaginal pulsing sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Other, specify: Vulva swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Other: Vaginal fullness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment and lack of subject participation/noncompliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04493333/Prot_SAP_000.pdf